CLINICAL TRIAL: NCT03695185
Title: A Multicenter, Single Arm, Open-label Study to Investigate the Efficacy and Safety of Ravagalimab (ABBV-323) in Subjects With Moderate to Severe Ulcerative Colitis Who Failed Prior Therapy
Brief Title: A Study to Investigate How Well Ravagalimab (ABBV-323) Works and How Safe it is in Participants With Moderate to Severe Ulcerative Colitis Who Failed Prior Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-722; 2018-000930-37 (EudraCT Number)
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Results first posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Ulcerative Colitis (UC); ABBV-323; Ravagalimab
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ravagalimab 600 mg/300 mg (Experimental): Participants received ravagalimab 600 mg intravenous (IV) at Week 0 followed by ravagalimab 300 mg subcutaneously (SC) at Weeks 2, 4, 6, 8, and 10 in a 12-week Induction Period. Participants who achieved clinical response per partial adapted Mayo score at Week 12 of the Induction Period entered the Maintenance Period to receive ravagalimab 300 mg SC every other week (EOW) from Week 12 through Week 102.
  Interventions: Drug: Ravagalimab 600 mg; Drug: Ravagalimab 300 mg

INTERVENTIONS:
Drug: Ravagalimab 600 mg — Ravagalimab 600 mg was administered intravenously (IV).
  Other Names: ABBV-323
Drug: Ravagalimab 300 mg — Ravagalimab 300 mg was administered subcutaneously (SC).
  Other Names: ABBV-323

SUMMARY:
Study M15-722 is a Phase 2a study to investigate the efficacy and safety of Ravagalimab (ABBV-323) in participants with moderate to severe UC who failed prior therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must voluntarily sign and date an informed consent, approved by an independent ethics committee (IEC)/institutional review board (IRB), prior to the initiation of any screening or study-specific procedures.
* Diagnosis of UC for at least 3 months prior to Baseline. Appropriate documentation of biopsy results consistent with the diagnosis of UC in the assessment of the Investigator, must be available.
* Participant meets the following disease activity criteria: Active UC with an Adapted Mayo score of 5 to 9 points and endoscopic subscore of 2 to 3 (confirmed by central review).
* History of inadequate response, loss of response, or intolerance to one or more of the approved biologic therapies: infliximab, adalimumab, golimumab, vedolizumab, and/or tofacitinib (Note: If tofacitinib was received in a clinical trial, subject must have received open-label drug).

Exclusion Criteria:

* Participant having an active, chronic, or recurrent infection that based on Investigator's clinical assessment makes the participant an unsuitable candidate for the study.
* Participant having any malignancy except for successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma or localized carcinoma in situ of the cervix.
* Participant with history of dysplasia of the gastrointestinal tract or evidence of dysplasia in any biopsy performed during the screening endoscopy other than completely removed low-grade dysplastic lesions.
* Laboratory values not meeting the following criteria : Serum aspartate transaminase (AST) and alanine transaminase (ALT) <= 2* upper limit of normal (ULN); Total white blood cell (WBC) count >= 3.0*10^9/L.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2022-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (34):
- United States (12):
  - Banner University Medical Cent /ID# 208392, Tucson, Arizona
  - Meridian Investigator Network /ID# 204646, Huntington Beach, California
  - Meridian Investigator Network /ID# 218568, Lakewood, California
  - TLC Clinical Research Inc /ID# 206626, Los Angeles, California
  - Orange County Institute of Gastroenterology and Endoscopy /ID# 207405, Mission Viejo, California
  - UC Davis Medical Center /ID# 209402, Sacramento, California
  - The University of Chicago DCAM /ID# 207086, Chicago, Illinois
  - Affinity Clinical Research /ID# 206211, Oak Brook, Illinois
  - Univ New Mexico /ID# 208817, Albuquerque, New Mexico
  - Penn Presbyterian Medical Center /ID# 206826, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center /ID# 204670, Nashville, Tennessee
  - Clinical Associates in Research Therapeutics of America, LLC /ID# 204689, San Antonio, Texas
- Mount Sinai Hospital /ID# 206180, Toronto, Ontario, Canada
- France (3):
  - Chu de Nice-Hopital L'Archet Ii /Id# 208131, Nice, Alpes-Maritimes
  - CHRU Nancy - Hôpitaux de Brabois /ID# 208133, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Hopital Beaujon /ID# 208129, Clichy, Île-de-France Region
- Germany (3):
  - Universitaetsklinikum Frankfurt /ID# 207569, Frankfurt am Main, Hesse
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 207571, Kiel, Schleswig-Holstein
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 207570, Berlin
- Hungary (2):
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont /ID# 221576, Szeged, Csongrád megye
  - Debreceni Egyetem Klinikai Kozpont /ID# 221952, Debrecen
- Italy (3):
  - University of Catanzaro /ID# 204546, Catanzaro, Calabria
  - Presidio Columbus-Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Un /ID# 204549, Rome, Roma
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 208504, Milan
- Netherlands (3):
  - Maastricht Universitair Medisch Centrum /ID# 204428, Maastricht
  - Franciscus Gasthuis & Vlietland /ID# 206976, Rotterdam
  - Elisabeth Tweesteden Ziekenhuis /ID# 206272, Tilburg
- South Korea (2):
  - Kyungpook National University Hospital /ID# 209912, Daegu
  - Yeungnam University Medical Center /ID# 210447, Daegu
- Spain (3):
  - Hospital Santa Creu i Sant Pau /ID# 213259, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 204504, Madrid
  - Hospital Universitario La Paz /ID# 210065, Madrid
- United Kingdom (2):
  - NHS Greater Glasgow and Clyde /ID# 206574, Glasgow, Scotland
  - Belfast Health and Social Care Trust /ID# 206744, Belfast

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 42 participants were enrolled in the Induction Period to receive ravagalimab 600 mg intravenously (IV) followed by ravagalimab 300 mg subcutaneously (SC) up to Week 12. Participants who completed the Induction Period and achieved clinical response per partial adapted Mayo score at Week 12 entered the Maintenance Period to receive ravagalimab 300 mg SC up to Week 102.
Pre-assignment Details: Prior to protocol version 4.0 this study was placebo-controlled. No participants were enrolled in the placebo group and therefore no results are presented for this arm.
Groups:
- Ravagalimab 600 mg/300 mg: Participants received ravagalimab 600 mg IV at Week 0 followed by ravagalimab 300 mg SC at Weeks 2, 4, 6, 8, and 10 in a 12-week Induction Period. Participants who achieved clinical response per partial adapted Mayo score at Week 12 of the Induction Period entered the Maintenance Period to receive ravagalimab 300 mg SC every other week (EOW) from Week 12 through Week 102.
Period: Induction Period (Week 0 to Week 12)
Arm/Group | Ravagalimab 600 mg/300 mg
Started | 42
Completed | 29
Not Completed | 13
Not completed — Adverse Event | 1
Not completed — Withdrew consent | 2
Not completed — Lack of Efficacy | 10
Period: Maintenance Period (Week 12 to Week 102)
Arm/Group | Ravagalimab 600 mg/300 mg
Started (Participants who completed the Induction Period and had a clinical response at Week 12 entered the Maintenance Period.) | 29
Completed | 1
Not Completed | 28
Not completed — Withdrew consent | 3
Not completed — Lack of Efficacy | 2
Not completed — Reason not specified | 23

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all enrolled participants who received at least 1 dose of ravagalimab and was used for all baseline and efficacy analyses.
Groups:
- Ravagalimab 600 mg/ 300 mg: Participants received ravagalimab 600 mg IV at Week 0 followed by ravagalimab 300 mg SC at Weeks 2, 4, 6, 8, and 10 in a 12-week Induction Period. Participants who achieved clinical response per partial adapted Mayo score at Week 12 of the Induction Period entered the Maintenance Period to receive ravagalimab 300 mg SC EOW from Week 12 through Week 102.
Arm/Group | Ravagalimab 600 mg/ 300 mg
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (14.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 39
  Race: Non-White | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Endoscopic Improvement During Induction Period
Description: Endoscopic Improvement is defined as Mayo endoscopic subscore of 0 or 1. Mayo endoscopic score is classified as 0=Normal or inactive disease; 1=Mild disease (erythema, decreased vascular pattern); 2=Moderate disease (marked erythema, absent vascular pattern, friability, erosions); 3=Severe disease (spontaneous bleeding, ulceration). Higher score indicates worsening of the disease. The number of responders is calculated based on the total number of participants and estimated response rate, rounding to a nearest whole integer.
Time Frame: At Week 8
Population: FAS included all enrolled participants who received at least 1 dose of ravagalimab. Data was reported only for the Induction Period.
Measure: Number; unit: percentage of participants
Groups:
- Ravagalimab 600 mg/300 mg: Participants received ravagalimab 600 mg IV at Week 0 followed by ravagalimab 300 mg SC at Weeks 2, 4, 6, 8, and 10 in a 12-week Induction Period.
Arm/Group | Ravagalimab 600 mg/300 mg
Number analyzed (Participants) | 42
percentage of participants | 18.0

2. Secondary Outcome: Percentage of Participants With Clinical Remission Per Adapted Mayo Score During Induction Period
Description: Clinical remission per Adapted Mayo score is defined as stool frequency subscore (SFS) <=1, and not greater than baseline, rectal bleeding subscore (RBS) = 0, and endoscopic subscore <=1. The Adapted Mayo Score is a composite score of UC disease activity based on the following 3 subscores: Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal), Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed), Endoscopic subscore confirmed by central reader, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration). The overall Adapted Mayo score ranges from 0 to 9 where higher scores represent more severe disease. The number of responders is calculated based on the total number of participants and estimated response rate, rounding to a nearest whole integer.
Time Frame: At Week 8
Population: FAS included all enrolled participants who received at least 1 dose of ravagalimab and was used for all baseline and efficacy analyses. Data was reported only for the Induction Period.
Measure: Number; unit: percentage of participants
Arm/Group | Ravagalimab 600 mg/300 mg
Number analyzed (Participants) | 42
percentage of participants | 9.5

3. Secondary Outcome: Percentage of Participants With Clinical Response Per Adapted Mayo Score During Induction Period
Description: Clinical response per Adapted Mayo score is defined as the decrease from Baseline >= 2 points and >= 30%, PLUS a decrease in RBS >=1 or an absolute RBS <=1. The Adapted Mayo Score is a composite score of UC disease activity based on the following 3 subscores: Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal), Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed), Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration). The overall Adapted Mayo score ranges from 0 to 9 with higher scores representing more severe disease. The number of responders is calculated based on the total number of participants and estimated response rate, rounding to a nearest whole integer.
Time Frame: At Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ravagalimab 600 mg/300 mg
Number analyzed (Participants) | 42
percentage of participants | 40.2

4. Secondary Outcome: Percentage of Participants With Clinical Response Per Partial Adapted Mayo Score
Description: Clinical response per Partial Adapted Mayo score is defined as decrease from baseline >=1 points and >=30%, PLUS a decrease in RBS >= 1 or an absolute RBS <=1. The Partial Adapted Mayo Score is a composite score of UC disease activity based on the following 2 subscores: SFS, scored from 0 (normal number of stools) to 3 (5 or more stools more than normal); RBS, scored from 0 (no blood seen) to 3 (blood alone passed). The overall Partial Adapted Mayo score ranges from 0 to 6 with higher scores representing more severe disease. The number of responders is calculated based on the total number of participants and estimated response rate, rounding to a nearest whole integer.
Time Frame: Up to Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ravagalimab 600 mg/300 mg
Number analyzed (Participants) | 42
percentage of participants | 57.1

5. Secondary Outcome: Percentage of Participants With Clinical Remission Per Full Mayo Score During Induction Period in Participants With a Full Mayo Score of 6 to 12 at Baseline
Description: Clinical Remission per full Mayo score is defined as Full Mayo score <=2 with no subscore > 1. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The FMS ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 4 subscores (stool frequency, rectal bleeding, endoscopy [confirmed by a central reader], and physician's global assessment), each of which ranges from 0 (normal) to 3 (severe disease). Endoscopies were assessed by a central reader. Negative changes indicate improvement. The number of responders is calculated based on the total number of participants and estimated response rate, rounding to the nearest whole integer.
Time Frame: At Week 8
Population: FAS included all enrolled participants who received at least 1 dose of ravagalimab. Overall number analysed is the number of participants available for analysis. Data was reported only for the Induction Period.
Measure: Number; unit: percentage of participants
Arm/Group | Ravagalimab 600 mg/300 mg
Number analyzed (Participants) | 40
percentage of participants | 7.5

6. Secondary Outcome: Percentage of Participants With Endoscopic Remission During Induction Period
Description: Endoscopic remission is defined as Mayo endoscopic subscore = 0. Endoscopies were assessed by a blinded central reader and scored according to the following scale: 0 = Normal or inactive disease; 1 = Mild disease (erythema, decreased vascular pattern); 2 = Moderate disease (marked erythema, lack of vascular pattern, any friability, erosions); 3 = Severe disease (spontaneous bleeding, ulceration). Higher score indicates worsening of the disease. The number of responders is calculated based on the total number of participants and estimated response rate, rounding to the nearest whole integer.
Time Frame: At Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Ravagalimab 600 mg/300 mg
Number analyzed (Participants) | 42
percentage of participants | 0.0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to safety follow up visit (up to approximately 116 weeks)
Description: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Induction Period: Ravagalimab 600 mg/300 mg: Participants received ravagalimab 600 mg IV at Week 0 followed by ravagalimab 300 mg SC at Weeks 2, 4, 6, 8, and 10 in a 12-week Induction Period.
- Maintenance Period: Ravagalimab 300 mg: Participants who achieved clinical response per partial adapted Mayo score at Week 12 of the Induction Period entered the Maintenance Period to receive ravagalimab 300 mg SC EOW from Week 12 through Week 102.
Arm/Group | Induction Period: Ravagalimab 600 mg/300 mg | Maintenance Period: Ravagalimab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/29
Serious Adverse Events (participants affected / at risk) | 2/42 | 2/29
Other Adverse Events (participants affected / at risk) | 15/42 | 19/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Period: Ravagalimab 600 mg/300 mg (N=42) | Maintenance Period: Ravagalimab 300 mg (N=29)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1) | 0 (0)
LARGE INTESTINE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PERIRECTAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Period: Ravagalimab 600 mg/300 mg (N=42) | Maintenance Period: Ravagalimab 300 mg (N=29)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 2 (2)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 2 (2)
HAEMORRHOIDS (Gastrointestinal disorders) | 3 (3) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 1 (1)
FATIGUE (General disorders) | 2 (7) | 3 (3)
PYREXIA (General disorders) | 2 (2) | 4 (5)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 2 (2)
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (7)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
HEADACHE (Nervous system disorders) | 2 (2) | 4 (4)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 3 (4)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT03695185/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT03695185/SAP_001.pdf